CLINICAL TRIAL: NCT04064281
Title: Effect of the Healthy Cantonese Diet on Cardiometabolic Syndrome in Chinese Adults
Brief Title: The Healthy Cantonese Diet on Cardiometabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CC-2019-03
Record Dates: First submitted 2019-08-12; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; High Blood Pressure; Hypertension; Hyperlipidemias; Hyperglycemia
Keywords: DASH; diet; trial; cardiovascular disease; blood pressure
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Hyperlipidemias; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: All subjects will enter 1-week run-in feeding period during which they will eat the control diet. After a 1-week run-in period, subjects will be randomly divided into the intervention group and the control group, stratified by gender. The two groups will eat their assigned diet for 4 consecutive weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the particularity of dietary intervention studies, it is hard to blind researchers and kitchen staff. Therefore, this trial only blinds subjects. In order to ensure blinding, they will be not told which group they have been assigned and the two groups will eat their assigned diet in different rooms. And outcomes assessors will also be blinded to the two diet groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the healthy Cantonese diet (Experimental): Based on the typical Cantonese diet, the healthy Cantonese diet is developed according to the DASH diet and the balanced dietary pattern of the Chinese Dietary Guidelines 2016. In this diet, the main nutrients, dietary fiber, sodium, calcium, magnesium and potassium are set to achieve the healthy goal. Compared with the typical Cantonese diet, the healthy Cantonese diet is increased in fruit, vegetables, low-fat dairy products, whole grains, nuts and seeds, and reduced in salt, oil and sweets.
  Interventions: Other: the healthy Cantonese diet
- the typical Cantonese diet (Placebo Comparator): The typical Cantonese diet is a diet of what many Cantonese eat. In this diet, the main nutrients, dietary fiber, sodium, calcium, magnesium and potassium are set at the average dietary intake levels in Guangdong.
  Interventions: Other: the typical Cantonese diet

INTERVENTIONS:
Other: the healthy Cantonese diet — After a 1-week run-in period, the intervention group will eat the healthy Cantonese diet for 4 consecutive weeks. Free meals will be provided 3 times a day (breakfast, lunch, dinner). The actually intake of every meal for all subjects will be recorded to estimate their nutrients intake. All subjects will be advised to avoid eating other food, but they should inform researchers of what they eat if they eat food that we will not provide.
  Arms: the healthy Cantonese diet
Other: the typical Cantonese diet — After a 1-week run-in period, the control group will still eat the typical Cantonese diet for 4 consecutive weeks. Free meals will be provided 3 times a day (breakfast, lunch, dinner). The actually intake of every meal for all subjects will be recorded to estimate their nutrients intake. All subjects will be advised to avoid eating other food, but they should inform researchers of what they eat if they eat food that we will not provide.
  Arms: the typical Cantonese diet

SUMMARY:
The DASH diet (Dietary Approaches to Stop Hypertension) have been proven to lower risk of cardiovascular diseases. But the DASH diet is inconsistent with Chinese dietary pattern. In this study, based on the typical Cantonese diet, the healthy Cantonese diet is developed according to the DASH diet and the balanced dietary pattern of the Chinese Dietary Guidelines 2016. The randomized control trial is designed to investigate whether the healthy Cantonese diet has benefit to blood pressure, blood lipid, blood glucose and other cardiometabolic biomarkers among adults with cardiometabolic syndrome in Guangdong, China.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-75 years old, male or female;
2. have lived in this community for the past six months, and have no plans to move out or go out in the next three months;
3. the systolic blood pressure is within 130-159mmHg regardless of medication.
4. maintaining the current medication (mainly drugs for hypertension, diabetes or hyperlipidemia) throughout the research period, with the category and dose unchanged;
5. the number of test meal consumed is no less than 18;
6. community feeding mode: eat a meal at least once a day at the research center (preferably lunch or dinner); or home delivery mode: upload meal pictures for three meals every day, and eat a meal and have physical examination at the research center at least once a week;
7. sign the informed consent form.

Exclusion Criteria:

1. fasting blood glucose ≥10.0mmol/L;
2. total cholesterol ≥7.2mmol/L;
3. injected inulin within a month;
4. unwilling or unable to change the original dietary pattern, or have special dietary needs (such as vegetarians);
5. alcoholism;
6. BMI ≥30kg/m^2, or losing weight currently;
7. have acute cardiovascular and cerebrovascular events occurred in the past six months;
8. have a history of chronic kidney disease, intestinal irritation or asthma;
9. women who have been/are preparing for pregnancy or lactation;
10. in combination with other serious diseases such as cancer, chronic heart failure, severe depression or other mental disorders, long-term bedridden or unable to move freely;
11. have a history of common food allergies (eggs, seafood, peanuts, etc.);
12. have undergone gastrointestinal surgery;
13. currently suffering from acute phase of diseases such as respiratory infections, fever, severe diarrhea;
14. have deaf-mutism, dementia, unable to communicate properly.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome score | before and after 4-week intervention
  Changes of metabolic syndrome score in healthy Cantonese diet compared with changes of typical Cantonese diet. Metabolic syndrome score will be derived by standardizing and then summing the following continuously distributed indices of adiposity (waist circumference) to create a z score: hypertension (the average of systolic blood pressure and diastolic blood pressure); hyperglycaemia (fasting plasma glucose); insulin resistance (fasting insulin); fasting HDL-cholesterol × -1; and fasting triacylglycerol z score.
Systolic blood pressure and diastolic blood pressure | before and after 4-week intervention
  Changes of systolic blood pressure and diastolic blood pressure in healthy Cantonese diet compared with changes of typical Cantonese diet. Blood pressure will be measured by trained investigator at baseline, week 1, week 2, week 3 and week 4, and systolic blood pressure and diastolic blood pressure will be recorded.
Blood lipid profile | before and after 4-week intervention
  Changes of blood lipid profile in healthy Cantonese diet compared with changes of typical Cantonese diet. Blood lipid profile (total cholesterol, TC; triglyceride, TG; LDL cholesterol, LDLc; HDL cholesterol, HDLc) will be tested by a validated biomedical analyses laboratory using vein serum at baseline and week 4.
Glucose metabolism | before and after 4-week intervention
  Changes of glucose metabolism in healthy Cantonese diet compared with changes of typical Cantonese diet. Glucose metabolism (fasting plasma glucose and fasting insulin) will be tested by a validated biomedical analyses laboratory using vein serum at baseline and week 4 and insulin resistance index (HOMA-IR) will be calculated by [fasting insulin (mU/L) × fasting plasma glucose (mmol/L) ]/22.5.

SECONDARY OUTCOMES:
Blood biochemical marker | before and after 4-week intervention
  Changes of blood biochemical marker in healthy Cantonese diet compared with changes of typical Cantonese diet. Blood biochemical marker (calcium, potassium, sodium, magnesium and phosphorus in mmol/L; uric acid in μmol/L) will be tested by a validated biomedical analyses laboratory using vein serum at baseline and week 4.
Urinary sodium and potassium | before and after 4-week intervention
  Changes of urinary sodium and potassium in healthy Cantonese diet compared with changes of typical Cantonese diet. Urinary sodium and potassium will be tested by a validated biomedical analyses laboratory using morning urine at baseline and week 4.
Intestinal microbiota composition | before and after 4-week intervention
  Changes of intestinal microbiota composition in healthy Cantonese diet compared with changes of typical Cantonese diet.
Gut microbial gene richness | before and after 4-week intervention
  Changes of gut microbial gene richness in healthy Cantonese diet compared with changes of typical Cantonese diet.
Inflammatory biomarkers | before and after 4-week intervention
  Changes of inflammatory biomarkers in healthy Cantonese diet compared with changes of typical Cantonese diet. Inflammatory biomarkers (CRP in mg/L; Tumor TNF-α and IL-6 in ng/L) will be tested by a validated biomedical analyses laboratory using vein serum at baseline and week 4.
Cardiopulmonary function | before and after 4-week intervention
  Changes of cardiopulmonary function in healthy Cantonese diet compared with changes of typical Cantonese diet. Cardiopulmonary function will be measured by cardiopulmonary exercise testing using CORTEX MetaLyzer 3B at baseline and week 4.
Endothelial function | before and after 4-week intervention
  Changes of endothelial function in healthy Cantonese diet compared with changes of typical Cantonese diet. Flow-mediated dilatation (FMD) will be assessed to evaluate endothelial function by using UNEX EF38G at baseline and week 4.
Body composition | before and after 4-week intervention
  Changes of body composition in healthy Cantonese diet compared with changes of typical Cantonese diet. Body composition will be tested by using dual energy X-ray absorptiometry at baseline and week 4.
Body mass index (BMI) | before and after 4-week intervention
  Height in meters and weight in kilograms will be combined to report body mass index (BMI) in kg/m^2.
Ratio of waist to hip circumference (WHR) | before and after 4-week intervention
  Waist circumference in centimeters and hip circumference in centimeters will be combined to report ratio of waist to hip circumference (WHR).